CLINICAL TRIAL: NCT04345172
Title: Lacrimal Dilator-Facilitated Incisionless Vs. Standard Sub-Tenon's Block: A Randomized, Prospective and Non-inferiority Comparative Study
Brief Title: Lacrimal Dilator-Facilitated vs Standard Sub-Tenon's Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Oya Yalcin Cok, Professor, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KA19/165
Record Dates: First submitted 2020-04-10; First posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: to Compare Lacrimal Dilator-facilitated Incisionless and Standard STB With Wescott Scissors
Keywords: sub-Tenon's block, lacrimal dilator, Wescott scissors, chemosis, subconjunctival haemorrhage

STUDY DESIGN:
Intervention Model Description: a randomized, prospective, non-inferiority comparative study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: triple blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a lacrimal dilator group (Group LD) (Active Comparator): The patients allocated to receive STB performed with a lacrimal dilator
  Interventions: Device: sub-Tenon's block with a lacrimal dilator group or a Wescott scissors
- a Wescott scissors (Group WS) (Active Comparator): The patients allocated to receive STB performed with a Wescott scissors
  Interventions: Device: sub-Tenon's block with a lacrimal dilator group or a Wescott scissors

INTERVENTIONS:
Device: sub-Tenon's block with a lacrimal dilator group or a Wescott scissors — Local anaesthetic eye drops were installed into the conjunctiva, followed by iodine 5% aqueous drops to the conjunctival sac for 3 minutes.19 An eye lid speculum was inserted.
  In group LD, the conjunctiva and Tenon's capsule were lifted together tightly with a blunt forceps like a tent in the inferonasal quadrant and a punctal dilatator (Castroviejo Lacrimal Dilatator, Katena Products, Inc, Denville, NJ, USA) was placed tangential to the globe creating a round and small hole at 5 mm posterior to limbus (Fig.1). The block was performed using smooth rounded tip, 19 G, 1 inch sub-Tenon's cannula (Visitec, Beaver-Visitec International Ltd, Warwickshire, UK).
  In Group WS, after lifting the conjunctiva and Tenon's capsule together with a blunt forceps, incision was performed with a blunt tip Westcott scissors in the inferonasal conjunctival at 5 mm posterior to limbus to expose sub-Tenon's space.

SUMMARY:
Standard sub-Tenon's block involves incision (dissection) of conjunctiva and Tenon's capsule with the help of blunt scissors and forceps, insertion of a blunt sub-Tenon's cannula under the Tenon's capsule and injection of local anaesthetic agent. This block is frequently associated with minor complications such as chemosis and subconjunctival haemorrhage. Different variations of incisionless sub-Tenon's block including the use of lacrimal dilator have been described to reduce minor complications and facilitate insertion of blunt cannula. Lacrimal dilator creates a small aperture in the conjunctiva and Tenon's capsule thus avoids incision. After ethics approval, patients undergoing elective cataract surgery were enrolled to receive sub-Tenon's block performed without incision with a lacrimal dilator (Group LD) or with incision using Wescott scissors and blunt forceps (Group WS). All patients received 3 mL 2% lidocaine without any adjuvant. No sedation was administered. Demographic of the patients, duration of the procedure, analgesia (pain), akinesia, duration of the procedure intraoperative chemosis, subconjunctival haemorrhage on the first postoperative day. We aimed to compare lacrimal dilator-facilitated and standard sub-Tenon's block effectiveness and incidence of chemosis and subconjunctival haemorrhage.

DETAILED DESCRIPTION:
The patients were randomly allocated to receive STB performed with a lacrimal dilator (Group LD) and with a Wescott scissors (Group WS). Randomization was ensured by sealed envelopes prepared according to a computer-generated table and the envelopes were opened by the operator just before the sub-Tenon's block.

Study protocol Local anaesthetic eye drops were installed into the conjunctiva, followed by iodine 5% aqueous drops to the conjunctival sac for 3 minutes.19 An eye lid speculum was inserted.

In group LD, the conjunctiva and Tenon's capsule were lifted together tightly with a blunt forceps like a tent in the inferonasal quadrant and a punctal dilatator was placed tangential to the globe creating a round and small hole at 5 mm posterior to limbus. The block was performed using smooth rounded tip, 19 G, 1 inch sub-Tenon's cannula .

In Group WS, after lifting the conjunctiva and Tenon's capsule together with a blunt forceps, incision was performed with a blunt tip Westcott scissors in the inferonasal conjunctival at 5 mm posterior to limbus to expose sub-Tenon's space. The block was performed with the above sub-Tenon's cannula.

All patients received lidocaine 2%, 3 mL without any adjuvant. No sedative was administered. All the blocks and surgeries were performed by the same investigator, but block evaluations were made by another investigator who was blinded to the technique used. All patients were discharged on the day of surgery.

The parameters recorded included demographic of the patients, duration of the procedure, analgesia (pain), akinesia, duration of the procedure intraoperative chemosis, subconjunctival haemorrhage on the first postoperative day. Analgesia was evaluated using a numeric rating scale for pain (0-10; 0 - no pain, 10 - the worst imaginable pain) immediately after the operation. Akinesia (ocular movements) were checked according to 4-primary gazes 10 minutes after STB. Chemosis and conjunctival haemorrhage (1st postoperative day) were assessed according to the number of quadrant or quadrants affected (superior nasal, superior temporal, inferior nasal, inferior temporal) using a 5-point scale (0-4; 0 - no for chemosis and haemorrhage, 4 for chemosis or haemorrhage in all 4 quadrants).

ELIGIBILITY:
Inclusion Criteria:

patients undergoing cataract surgery by phacoemulsification and intraocular lens implantation

Exclusion Criteria:

allergy to lidocaine, history of previous retinal and strabismus surgery, bleeding disorders and oral anticoagulant use, presence of glaucoma or high IOP, thick pterygia, any pathological condition that conjunctiva and Tenon's capsule cannot be lifted away from the sclera

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
chemosis | 10 minutes after intervention
  swelling of the conjunctiva

SECONDARY OUTCOMES:
subconjunctival haemorrhage | on the postoperative first day
  haemorrhage due to tearing or severing of blood vessels during dissection and injection

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Adana Research and Training Center, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
This will be decided according to the content of the request